CLINICAL TRIAL: NCT05944055
Title: Is 25OHD Overdoses Before 36 Weeks Corrected Age an Independant Risk Factor of Bronchopulmonary Dysplasia or Death ?
Brief Title: 25OH Vitamin D Overdoses and Risk of Bronchopulmonary Dysplasia or Death
Acronym: 25OHVDORBPDD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0244
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Bronchopulmonary Dysplasia; Vitamin D Overdose
Keywords: vitamin D; Overdoses; Bronchopulmonary Dysplasia; Preterm infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Drug Overdose | interventions — Death Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overdose: Preterm born before 31 weeks of gestation with at least a 25OH-D measure above 120nmol/L before 36 weeks corrected age and no determination below 50nmol/L. Of note, 25OH-D determinations are routinely performed each month from the first month of life during the NICU hospitalization
  Interventions: Biological: Is 25 OH vitamin D overdose a risk factor of bronchopulmonary dysplasia or death ?
- Control: Preterm infants born before 31 weeks of gestation, who presented with a 25OH-D between 50 and 120nmol/L for all the 25OH-D measures during their hospitalization in the NICU setting.
  Of note, 25OH-D determinations are routinely performed each month from the first month of life during the NICU hospitalization
  Interventions: Biological: Is 25 OH vitamin D overdose a risk factor of bronchopulmonary dysplasia or death ?

INTERVENTIONS:
Biological: Is 25 OH vitamin D overdose a risk factor of bronchopulmonary dysplasia or death ? — Vitamin D overdose is frequent among preterm infants receiving the current supplementation (Mauras 2022, Kołodziejczyk-Nowotarska 2021). In our NICU, the protocol was to daily administrate 55 UI vitamin D during parenteral nutrition then 1000 UI during enteral nutrition for babies weighing more than 1000 g and 1200UI during enteral nutrition for babies weighing less than 1000 g. The dosage was adapted each month after a plasmatic measure of 25OH-D in order to maintain 25OH-D between 50 nmol/L and 120 nmol/L.

SUMMARY:
Several studies have demonstrated that vitamin D deficiency at birth is a risk factor of bronchopulmonary dysplasia. However, in an animal model of bronchopulmonary dysplasia vitamin D overdose has also been associated with an increased mortality and an increased lung injury. Such vitamin D overdose has been frequently reported in hospitalized neonates receiving the current supplementation.

The hypothesis is that vitamin D overdose is an independent risk factor of bronchopulmonary dysplasia or death among infants born below 31 weeks gestational age excluding infants with vitamin D deficiency.

This retrospective cohort study will include all infants born before 31 weeks of gestation (WG), who were hospitalized in a tertiary neonatal intensive care unit (NICU) during at least 10 days, for who at least one 25OH vitamin D determination was performed before 36 WG corrected age and whose parents are not opposed to the study. A descriptive analysis of the cohort depending on the occurrence of vitamin D overdose will be performed. A multivariate analysis will determine if vitamin D overdose is an independent risk factor of bronchopulmonary dysplasia or death among preterm infants, adjusting on the covariates known to be associated with bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria * :
* Infant born before 31 weeks of gestation.
* hospitalized in the NICU during at least 10 days
* with at least a 25OH-D determination available before 36 weeks corrected age

Exclusion Criteria:

-Infant with at least a 25OH-D below 50 nmol/L

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants hospitalized in the NICU at Hôpital Femme Mère Enfant, Bron, France. With a measure of 25OHD each month from the first month of life, as routinely recommended in this NICU.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia or death | The outcome will be assessed at 36 weeks corrected age.
  Bronchopulmonary dysplasia is defined as any respiratory support or oxygen requirement at 36 weeks corrected age.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France